CLINICAL TRIAL: NCT03227497
Title: Investigation of Health Effects of Dietary Intake of Whole Walnuts in Adult Subjects Under Low Cardiovascular Risk Towards Established and Molecular Cardiovascular Risk Factors
Brief Title: Dietary Intake of Whole Walnuts in Adult Subjects Under Low Cardiovascular Risk
Acronym: FitALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Collaborators: Centre of Research Excellence in Nutrition and Metabolism (Unknown)
Responsible Party: Principal Investigator, Manja Zec, Dr, University of Belgrade
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EO120/2017
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Cardiovascular Risk Factor; Metabolic Syndrome; Hypertension
Keywords: Blood Pressure; Cholesterol; Triglycerides; Walnuts
MeSH Terms: conditions — Metabolic Syndrome; Hypertension

STUDY DESIGN:
Intervention Model Description: This study is a randomized, cross-over, controlled, 5-week nutritional intervention, investigating health effects of dietary intake of whole walnuts, as a replacement meal within habitual diet and lifestyle.
  At the beginning of the study, half of the study subjects are randomly assigned to a treatment arm with walnut consumption, or control arm without study intervention. Treatment arm considers consumption of pre-packed 56 g of whole walnuts daily, as a replacement meal. After 5 weeks, study subjects are crossed, for additional 5 weeks. At the beginning of the study, all subjects are instructed to continue with their habitual diet and physical activity during the study period of 10 weeks.
Masking Description: Independent researcher will perform statistical analyses, without prior knowledge on study treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walnut (Active Comparator): At the beginning of the study, subjects are randomly assigned to receive either intervention treatment (whole walnuts) or no treatment (control arm).
  Treatment arm includes 56 g of whole walnuts daily.
  Interventions: Dietary Supplement: Whole Walnuts
- Control (No Intervention): At the beginning of the study, subjects are randomly assigned to receive either intervention treatment (whole walnuts) or no treatment (control arm).

INTERVENTIONS:
Dietary Supplement: Whole Walnuts — Intervention arm includes whole walnuts taken as dietary replacement meal during the day, and between breakfast and lunch, and/or lunch and dinner. Importantly, none of the main meals, including breakfast, lunch and dinner are to be replaced by study intervention, and the study subjects are instructed to do so. Walnuts are provided with the same producer at the Belgrade market.
  Arms: Walnut

SUMMARY:
This cross-over study investigates health effects of dietary intake of whole walnuts towards cardiovascular risk factors in adults under low cardiovascular risk.

Investigators hypothesize that daily intake of whole nuts as a replacement meal, would improve cardiovascular risk factors, including traditional risk factors and molecular biomarkers.

The participants are randomly assigned to receive either study treatment, or no treatment, and are crossed after five weeks.

The study subjects are instructed to continue with their habitual diet and physical activity.

DETAILED DESCRIPTION:
Recent literature data raise important questions on the beneficial effect of dietary fats. Dietary intake of nuts, although with high caloric burden, is however characterized with high intake of fatty acids with known beneficial health effects. Those fatty acids include mono- (MUFA) and polyunsaturated fatty acids (PUFA), to whom beneficial health effects are ascribed.

Among nuts, walnuts are characterized with comparatively high levels of MUFA and PUFA, especially content of alpha-linolenic PUFA, considered essential fatty acid, since not synthesized endogenously in humans. Dietary intake of alpha-linolenic acid is shown to be inversely related with cardiovascular risk factors, both in interventional studies and epidemiological cohorts. Molecular background of alpha-linolenic actions is bidirectional, and includes the action itself, as well as beneficial endogenous conversion towards long-chain fatty acids, including eicosapentaenoic and docosahexaenoic fatty acid.

Although high caloric intake is indicated with intake of walnuts, literature data suggest that consumption of walnuts does not increase body weight.

Dietary intake of walnuts has been shown to decrease cholesterol fractions, triglycerides and apolipoproteins in adult population. Also, consumption of walnuts was associated with decrease in blood pressure.

The study design is cross-over, controlled, randomized nutritional intervention. The participants are randomly assigned to receive either study treatment, or no treatment, and are crossed after five weeks.

The study subjects are instructed to continue with their habitual diet and physical activity. Additionally, study subjects are instructed to avoid walnuts and nuts other then study treatment, during the complete study period of 10 weeks.

Sample size calculation was conducted by use of online calculators, and was based on the low density lipoprotein (LDL) cholesterol. Namely, in order to achieve decrease in 0.5 mmol/L, in a sample with projected standard deviation of 0.7 mmol/L, and type I and II errors being 0.2 and 0.05, respectively, 62 subjects are needed.

ELIGIBILITY:
Inclusion Criteria:

Presence of at least one of the following criteria, formerly assessed through routine medical examination:

* dyslipidemia, defined as the presence of either: elevated total cholesterol (>5.2 mmoL/L), and/or elevated LDL-cholesterol (>3.4 mmoL/L), and/or elevated triglycerides (>1.7 mmoL/L), and/or decreased HDL-cholesterol (<1.6 mmoL/L)
* elevated blood pressure (systolic/diastolic ≥120/80 mmHg), or regular anti-hypertension therapy

Exclusion Criteria:

* presence of allergy on any nuts
* presence of any chronic disease, excluding following conditions: hypertension and diabetes mellitus type 2
* smoking
* statin therapy
* pregnancy and/or lactation

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Changes in LDL-cholesterol | Baseline, 5 weeks, 10 weeks
  Changes in LDL-cholesterol measured by clinical bio-analyzer from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in Systolic Blood Pressure | Baseline, 5 weeks, 10 weeks
  Changes in Systolic Blood Pressure, from baseline to endpoint, measured office-based at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in Diastolic Blood Pressure | Baseline, 5 weeks, 10 weeks
  Changes in Diastolic Blood Pressure from baseline to endpoint, measured office-based at the following timepoints: 0 (baseline), 5 and 10 weeks.

SECONDARY OUTCOMES:
Changes in HDL-cholesterol | Baseline, 5 weeks, 10 weeks
  Changes in HDL-cholesterol measured by clinical bio-analyzer from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in total cholesterol | Baseline, 5 weeks, 10 weeks
  Changes in total cholesterol measured by clinical bio-analyzer from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in triglycerides | Baseline, 5 weeks, 10 weeks
  Changes in triglycerides measured by clinical bio-analyzer from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in glucose metabolism biomarkers | Baseline, 5 weeks, 10 weeks
  Changes in glucose biomarkers measured by clinical bio-analyzer from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in renal function parameters | Baseline, 5 weeks, 10 weeks
  Changes in renal function parameters measured by clinical bio-analyzer from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in liver function parameters | Baseline, 5 weeks, 10 weeks
  Changes in liver function parameters measured by clinical bio-analyzer from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in body weight | Baseline, 5 weeks, 10 weeks
  Changes in body weight measured by bio-impedance analyzer, from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in waist circumference | Baseline, 5 weeks, 10 weeks
  Changes in waist circumference, from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in percent of total body fat | Baseline, 5 weeks, 10 weeks
  Changes in percent of total body fat measured by bio-impedance analyzer, from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
Level of Physical Activity | Baseline
  Level of physical activity is assessed by use of standardized Physical Activity Questionnaire.
Psychological parameters | 5 weeks
  Psychological parameters are assessed by use of standardized questionnaire for self-assessment of psychological implications of daily activities related to cardiovascular health .
Changes in hematological parameters | Baseline, 5 weeks, 10 weeks
  Changes in hematological, from baseline to endpoint, measured by hematological clinical analyzer at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in number of leukocyte cells | Baseline, 5 weeks, 10 weeks
  Changes in number of leukocyte cells, from baseline to endpoint, measured by hematological clinical analyzer at the following timepoints: 0 (baseline), 5 and 10 weeks.
Changes in total caloric intake | Baseline, 5 weeks, 10 weeks
  Changes in total caloric intake, from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
  Total caloric intake is measured by use of standardized dietary questionnaire namely 24-hour Dietary Recall.
Changes in caloric intake of fats | Baseline, 5 weeks, 10 weeks
  Changes in caloric intake of fats, from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
  The caloric intake is measured by use of standardized dietary questionnaire, namely 24-hour Dietary Recall.
Changes in caloric intake of carbohydrates | Baseline, 5 weeks, 10 weeks
  Changes in caloric intake of carbohydrates, from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
  The caloric intake is measured by use of standardized dietary questionnaire, namely 24-hour Dietary Recall.
Changes in caloric intake of vitamin D | Baseline, 5 weeks, 10 weeks
  Changes in caloric intake of vitamin D, from baseline to endpoint, measured at the following timepoints: 0 (baseline), 5 and 10 weeks.
  The caloric intake is measured by use of standardized dietary questionnaire, namely 24-hour Dietary Recall.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Glibetic, Prof, Principal Investigator — Center of Research Excellence in Nutrition and Metabolism, Institute for Medical Resaerch
Locations (1):
- Center of Research Excellence in Nutrition and Metabolism, Institute for Medical Research, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No